CLINICAL TRIAL: NCT07352527
Title: New Clinical Decision Support Score Based on Steroid Hormone Profiling in the Diagnosis of Adrenal Adenomas With Moderate Autonomous Cortisol Secretion or MACS
Brief Title: New Clinical Decision Support Score Based on Steroid Hormone Profiling in the Diagnosis of MACS
Acronym: MACSCORE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/28
Record Dates: First submitted 2025-09-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Endocrine Disease
Keywords: Mild autonomous cortisol secreting adrenocortical adenoma; steroid hormone profiling; steroid metabolome; LC-MS/MS
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MACS group: Mild autonomous cortisol-secreting adenoma group must at least have two elevated DST1mg (Cortisol > 50 nmol/L or 1.8 µg/dL) and a plasma ACTH level ≤ 20 pg/mL
- ANS group: Non-secreting adenoma must have a normal DST1mg (Cortisol ≤ 50 nmol/L or 1.8 µg/dL).
- Control group: Control group is patients followed in the endocrinology department, free of any known adrenal pathology and with a DST1mg test < 50nmol/L and matched for age and sex to patients in groups 1 and 2.

SUMMARY:
The recent development of quantitative steroid metabolome profiling could be of interest for the positive diagnosis of mild autonomous cortisol-secreting adenoma (MACS). The aim of the study is to develop a predictive model of MACS status or non-secreting adenoma (NSA) based on a panel of 19 serum steroids and three clinico-biological parameters (body mass index or BMI, fasting glycaemia, blood pressure) and to estimate its performance for the diagnosis of MACS in a cohort of patients followed in the endocrinology department of Bordeaux University Hospital.

DETAILED DESCRIPTION:
Steroid assays are a central element in the aetiological diagnosis of adrenal tumors, but they are still limited to single assays (e.g. cortisol in Cushing's syndrome, aldosterone in primary hyperaldosteronism, etc.) which only partially reflect the endocrine disturbances caused by adrenal pathologies. The recent development of quantitative profiling of the circulating steroidome could lead to a reconsideration of the role of these single steroid assays in endocrinology. This involves simultaneously measuring of multiple steroids from a single blood or urine sample using liquid chromatography-mass spectrometry (LC-MS/MS). The steroid fingerprint obtained enables adrenal masses to be better characterised. Using machine learning methods, a predictive model of MACS status or NSA based on a panel of 19 serum steroids measured by LC-MS/MS and three clinico-biological parameters (body mass index or BMI, fasting glycaemia, blood pressure) will be develop. The blood sample used for the steroid assay will be taken at inclusion during a blood test carried out as part of routine care. Clinical, biological and morphological data obtained during the 24 months of study follow-up and as part of routine care will be collected retrospectively. All assays will be carried out in the hormonology laboratory of Bordeaux University Hospital (BUH) by LC-MS/MS. The development of the MACS/ANS status prediction model will be carried out by the BUH Methodological Support Unit for Clinical and Epidemiological Research (USMR). The performance and prognostic value of this new tool will be estimated in a cohort of patients followed in the BUH endocrinology department.

ELIGIBILITY:
Inclusion Criteria:

MACS and ANS group:

* 18 years ≤ Age
* Patient with one or more unilateral or bilateral adrenal nodules with spontaneous density < 20 HU on CT and major axis ≥ 1 cm and without associated overt pathological hormonal secretion.
* Patient with one or more uni or bilateral adrenal nodules not meeting the above density criteria but without malignancy criteria and stable in size on imaging after at least 6 months of follow-up and without associated overt pathological hormone secretion.
* Written consent of the patient for his participation in the research (at the latest on the day of inclusion and before any examination required by the research).
* Subject affiliated to or benefiting from a social security scheme.

Diagnostic criteria (determined after blood sampling) for continuation of the study:

MACS group:

* At least two elevated DST1mg (Cortisol > 50 nmol/L or 1.8 µg/dL) AND
* a plasma ACTH level ≤ 20 pg/mL

ANS group:

- Normal DST1mg (Cortisol ≤ 50 nmol/L or 1.8 µg/dL). The definition criteria for MACS and ANS were based on the latest recommandations of learned societies.

Controls group:

* patients followed in the endocrinology department, free of any known adrenal pathology and with a DST1mg test < 50nmol/L.
* matched for age and sex to patients in groups 1 and 2.

Non -inclusion criteria:

* Adrenal incidentaloma < 1 cm in size.
* Use of exogenous corticosteroids, whether systemic or local (inhaled, eye and ear drops, ophthalmic ointment, topical skin products, joint infiltration) in the 6 months prior to the trial, and drugs that interfere with the metabolism of dexamethasone.
* Pregnant women.
* Patients with any other life-threatening condition.
* Patients with an intercurrent pathology at the time of blood sampling (fever, COVID infection, influenza....).
* Urinary free cortisol (UFC) > at the limit of laboratory normality.
* Patients under court protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The feasibility of the project is ensured by active and ongoing collaboration between:
  * The endocrinology department at Bordeaux University Hospital, which has recognized expertise in adrenal disorders, particularly MACS (participation in drafting European recommendations on adrenal incidentalomas, reference centers for rare adrenal diseases). It has strong potential for recruiting patients monitored for adrenal disorders throughout the Nouvelle-Aquitaine region.
  * The hormone department at Bordeaux University Hospital, itself a reference center for LC-MS/MS steroid dosing and active in research projects on this topic.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the prediction model's performance | 18 months after inclusion
  Performance will be evaluated by internal validation using bootstrap sampling of 1,000 samples, and by the discrimination of the model by the ROC curve.

SECONDARY OUTCOMES:
Correlation between blood steroid levels and blood pressure | 18 months after inclusion
  The correlation between blood steroid levels and blood pressure will be evaluated in patients with MACS by correlating blood steroid concentrations and blood pressure thanks to ambulatory blood pressure monitoring which record 3 measurements during 3 consecutive days, and calculate after an average systolic and diastolic BP
Correlation between blood steroid levels and Body Mass Index | 18 months after inclusion day
  The correlation between blood steroid levels and Body Mass Index (BMI) will be evaluated in patients with MACS by correlating blood steroid concentrations obtain by dosages and calculated BMI (weight/size²).
Correlation between blood steroid levels and carbohydrate tolerance | 18 months after inclusoin day
  The correlation between blood steroid levels and carbohydrate tolerance will be evaluated in patients with MACS by correlating blood steroid concentrations and fasting blood glucose dosage, Hba1c, blood glucose levels 2 hours after glucose tolerance test.
Correlation between blood steroid levels and bone mineral density | 18 months after inclusion day
  The correlation between blood steroid levels and bone mineral density will be evaluated in patients with MACS by correlating blood steroid concentrations and bone mineral density thanks to bone densitometry.
Correlation between blood steroid levels and bone architecture | 18 months after inclusion day
  The correlation between blood steroid levels and bone architecture will be evaluated in patients with MACS by correlating blood steroid concentrations and bone architecture thanks to Trabecular Bone Score (TBS).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Haut-Lévêque, Pessac, France

IPD SHARING:
Plan to Share IPD: No